CLINICAL TRIAL: NCT00003945
Title: A Randomized Phase III Study of Cisplatin Versus Cisplatin Plus Topotecan Versus MVAC in Stage IVB, Recurrent or Persistent Squamous Cell Carcinoma of the Cervix
Brief Title: Comparison of Three Chemotherapy Regimens in Treating Patients With Stage IVB, Recurrent, or Persistent Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067138; GOG-0179; ECOG-G0179
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2004-09

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; stage IVB cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Topotecan

INTERVENTIONS:
Drug: cisplatin
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective for cervical cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of three different chemotherapy regimens in treating patients with stage IVB, recurrent, or persistent cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rate and survival of patients with stage IVB, recurrent, or persistent carcinoma of the cervix treated with cisplatin only vs cisplatin plus topotecan vs methotrexate, vinblastine, doxorubicin, and cisplatin (MVAC). (Arm III (MVAC) closed to accrual effective 07/23/2001.)
* Compare the toxic effects of these regimens in this patient population.
* Compare health-related quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to GOG performance status. Patients are randomized to one of three treatment arms. (Arm III closed to accrual effective 07/23/2001.)

* Arm I: Patients receive cisplatin IV once every 21 days.
* Arm II:Patients receive topotecan IV over 30 minutes on days 1-3 and cisplatin IV (beginning after topotecan infusion) on day 1. Courses repeat every 21 days.
* Arm III:Patients receive methotrexate IV on days 1, 15, and 22, vinblastine IV on days 2, 15, and 22, and doxorubicin IV and cisplatin IV on day 2. Courses repeat every 28 days. (Arm III closed to accrual effective 07/23/2001.) Treatment in all arms continues for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. (Arm III closed to accrual effective 07/23/2001.)

Quality of life is assessed before randomization, before course 2, before course 5 (arms I and II), before course 4 (arm III), and at 9 months. (Arm III closed to accrual effective 07/23/2001.)

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 400 patients (133 per treatment arm) will be accrued for this study within 2 years. (Arm III closed to accrual effective 07/23/2001.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IVB, recurrent, or persistent carcinoma of the cervix that is not amenable to curative treatment with surgery and/or radiotherapy

  * Eligible subtypes:

    * Squamous cell carcinoma
    * Adenosquamous carcinoma
    * Adenocarcinoma
* Measurable disease by physical examination, radiography, CT scan, or MRI

  * Measurable disease by CT scan/MRI without biopsy confirmation allowed if lesions are at least 3 cm and well defined
* No craniospinal metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Alkaline phosphatase no greater than 3 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL
* No bilateral hydronephrosis that cannot be alleviated by ureteral stents or percutaneous drainage

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No clinically significant infection
* No other prior invasive malignancy within the past 5 years except nonmelanoma skin cancer
* Body surface area no greater than 2.0 m^2

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 6 weeks since prior chemoradiotherapy and recovered
* No prior chemotherapy except when used concurrently with radiotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* See Chemotherapy
* At least 3 weeks since prior radiotherapy only and recovered

Surgery:

* Recovered from prior surgery

Other:

* No prior anticancer treatment that would preclude study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 1999-06; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry J. Long, MD, Study Chair — Mayo Clinic; Higinia R. Cardenes, MD, PhD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (11):
- United States (8):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center-Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Background] Chase DM, Huang HQ, Wenzel L, Cella D, McQuellon R, Long HJ, Moore DH, Monk BJ. Quality of life and survival in advanced cervical cancer: a Gynecologic Oncology Group study. Gynecol Oncol. 2012 May;125(2):315-9. doi: 10.1016/j.ygyno.2012.01.047. Epub 2012 Feb 1. PMID 22307062
- [Background] Moore DH, Tian C, Monk BJ, Long HJ, Omura GA, Bloss JD. Prognostic factors for response to cisplatin-based chemotherapy in advanced cervical carcinoma: a Gynecologic Oncology Group Study. Gynecol Oncol. 2010 Jan;116(1):44-9. doi: 10.1016/j.ygyno.2009.09.006. Epub 2009 Oct 22. PMID 19853287
- [Background] Paton F, Paulden M, Saramago P, Manca A, Misso K, Palmer S, Eastwood A. Topotecan for the treatment of recurrent and stage IVB carcinoma of the cervix. Health Technol Assess. 2010 May;14 Suppl 1:55-62. doi: 10.3310/hta14Suppl1/08. PMID 20507804
- [Background] Plaxe SC, Brooks SE, Tian C, Bloss JD, Moore DH, Long HJ. Influence of race on tolerance of platinum-based chemotherapy and clinical outcomes in women with advanced and recurrent cervical cancer: a pooled analysis of 3 Gynecologic Oncology Group studies. Am J Obstet Gynecol. 2008 Nov;199(5):539.e1-6. doi: 10.1016/j.ajog.2008.04.038. Epub 2008 Jun 20. PMID 18565487
- [Background] Moore DH, Tian C, Monk BJ, et al.: Factors predictive of response to cisplatin-based chemotherapy in stage IVB persistent or recurrent cervical carcinoma: a multivariate analysis of three Gynecologic Oncology Group trials. [Abstract] J Clin Oncol 25 (Suppl 18): A-5534, 282s, 2007.
- [Background] Tewari KS, Monk BJ. Gynecologic oncology group trials of chemotherapy for metastatic and recurrent cervical cancer. Curr Oncol Rep. 2005 Nov;7(6):419-34. doi: 10.1007/s11912-005-0007-z. PMID 16221379
- [Result] Long HJ 3rd, Monk BJ, Huang HQ, Grendys EC Jr, McMeekin DS, Sorosky J, Miller DS, Eaton LA, Fiorica JV; Gynecologic Oncology Group. Clinical results and quality of life analysis for the MVAC combination (methotrexate, vinblastine, doxorubicin, and cisplatin) in carcinoma of the uterine cervix: A Gynecologic Oncology Group study. Gynecol Oncol. 2006 Mar;100(3):537-43. doi: 10.1016/j.ygyno.2005.09.023. Epub 2005 Oct 10. PMID 16216315
- [Result] Long HJ 3rd, Bundy BN, Grendys EC Jr, Benda JA, McMeekin DS, Sorosky J, Miller DS, Eaton LA, Fiorica JV; Gynecologic Oncology Group Study. Randomized phase III trial of cisplatin with or without topotecan in carcinoma of the uterine cervix: a Gynecologic Oncology Group Study. J Clin Oncol. 2005 Jul 20;23(21):4626-33. doi: 10.1200/JCO.2005.10.021. Epub 2005 May 23. PMID 15911865
- [Result] Monk BJ, Huang HQ, Cella D, Long HJ 3rd; Gynecologic Oncology Group Study. Quality of life outcomes from a randomized phase III trial of cisplatin with or without topotecan in advanced carcinoma of the cervix: a Gynecologic Oncology Group Study. J Clin Oncol. 2005 Jul 20;23(21):4617-25. doi: 10.1200/JCO.2005.10.522. Epub 2005 May 23. PMID 15911864
- [Result] Grendys EC Jr, Long HJ, Bundy BN, et al.: Randomized phase III trial of cisplatin vs cisplatin plus topotecan vs the combination of methotrexate, vinblastine, doxorubicin, and cisplatin (MVAC) in stage IVB, recurrent or persistent carcinoma of the uterine cervix: a Gynecologic Oncology Group study. [Abstract] Int J Gynecol Cancer 14 (Suppl 1): A-039, 12, 2004.
- [Result] Monk BJ, Huang H, Cella D, et al.: Quality of life outcomes from GOG 179: a phase III trial of cisplatin vs cisplatin/topotecan in recurrent or persistent carcinoma of the cervix. [Abstract] Int J Gynecol Cancer 14 (Suppl 1): A-142, 42, 2004.